CLINICAL TRIAL: NCT06411275
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study to Evaluate the Efficacy and Safety of HTD1801 in Patients With Type 2 Diabetes Mellitus (T2DM) Inadequately Controlled With Diet and Exercise
Brief Title: A Phase 2 Study of Berberine Ursodeoxycholate (HTD1801) in Patients With Type 2 Diabetes Inadequately Controlled With Diet and Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Collaborators: Shenzhen HighTide Biopharmaceutical Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTD1801.PCT103
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HTD1801 500 mg (Experimental): Administered orally twice daily (BID)
  Interventions: Drug: HTD1801
- HTD1801 1000 mg (Experimental): Administered orally BID
  Interventions: Drug: HTD1801
- Placebo (Placebo Comparator): Administered orally BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTD1801 — HTD1801 administered orally BID as two capsules
  Other Names: berberine ursodeoxycholate
  Arms: HTD1801 500 mg
Drug: Placebo — Matching placebo administered orally BID as two to four capsules
  Arms: Placebo
Drug: HTD1801 — HTD1801 administered orally BID as four capsules
  Other Names: berberine ursodeoxycholate
  Arms: HTD1801 1000 mg

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of berberine ursodeoxycholate (HTD1801) compared to placebo in patients with type 2 diabetes inadequately controlled with diet and exercise alone.

DETAILED DESCRIPTION:
This Phase 2 randomized, double-blind, placebo-controlled trial will evaluate the efficacy and safety of HTD1801 compared to placebo after 12-weeks of treatment.

To ensure stabilization of glycemic control, eligible patients will first participate in a 4-week single-blind run-in period where investigators will provide guidance on lifestyle modification, concomitant medications, and procedures for self-monitoring of blood glucose. Following this period, patient eligibility will be reassessed. Eligible patients will be randomized 1:1:1 to receive HTD1801 500 mg twice daily (BID), HTD1801 1000 mg BID, or placebo BID.

ELIGIBILITY:
Key Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus according to the 1999 World Health Organization (WHO) criteria
* Have followed dietary and exercise interventions for at least 8 weeks prior to screening
* Have HbA1c ≥7.5% to ≤11.0% (screening) and ≥7.0% to ≤10.5% (pre-randomization)
* Have fasting plasma glucose <13.9 mmol/L (screening and pre-randomization)
* Have a body mass index ≥18 kg/m^2 to ≤40 kg/m^2

Key Exclusion Criteria:

* Have type 1 diabetes mellitus or specific type of diabetes mellitus (pancreatic injury-induced diabetes mellitus, diabetes mellitus caused by Cushing's syndrome or acromegaly, etc.)
* Have had diabetic ketoacidosis or hyperglycemic hyperosmolar state within 6 months prior to screening
* Have had 2 or more Grade 3 hypoglycemic events within 12 months prior to screening
* Have unstable or treatment-requiring proliferative retinopathy or macular degeneration, severe diabetic neuropathy, diabetic foot, or intermittent claudication within 6 months prior to screening
* Have been taking any weight loss medication or dietary supplement, have participated in a weight loss program, or have adhered to a special diet within 4 weeks prior to screening
* Have continuously used insulin or an insulin analogue for more than 14 days within 12 months prior to screening
* Have used 2 or more classes of hypoglycemic medications for more than 8 weeks within 12 months prior to screening
* Have used any glucose-modifying medications within 8 weeks prior to screening
* Have had weight gain or loss ≥5% from screening to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c | 12 Weeks
  Mean change in HbA1c from baseline to Week 12

SECONDARY OUTCOMES:
Mean change in fasting plasma glucose | 12 Weeks
  Mean change in fasting plasma glucose from baseline to Week 12
Proportion of patients achieving HbA1c <7.0% | 12 Weeks
  Proportion of patients achieving HbA1c <7.0% after 12 weeks of treatment
Proportion of patients achieving HbA1c <6.5% | 12 Weeks
  Proportion of patients achieving HbA1c <6.5% after 12 weeks of treatment
Mean change in postprandial glucose | 12 Weeks
  Mean change in postprandial glucose from baseline to Week 12
Mean change in low-density lipoprotein cholesterol (LDL-C) | 12 Weeks
  Mean change in LDL-C from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Kui Liu, Study Director — Shenzhen HighTide Biopharmaceutical Ltd.
Locations (14):
- China (14):
  - Peking University People's Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Huizhou Municipal Central Hospital, Huizhou
  - Jinan Central Hospital, Jinan
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Nanjing First Hospital, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - Sir Run Run Hospital Nanjing Medical University, Nanjing
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Yan'an University Affiliated Hospital, Yanan
  - Affiliated Hospital of Jiangsu University, Zhenjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji L, Ma J, Ma Y, Cheng Z, Gan S, Yuan G, Liu D, Li S, Liu Y, Xue X, Bai J, Wang K, Cai H, Li S, Liu K, Yu M, Liu L. Berberine Ursodeoxycholate for the Treatment of Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e2462185. doi: 10.1001/jamanetworkopen.2024.62185. PMID 40029660